CLINICAL TRIAL: NCT03511300
Title: Ready Set Goal: A Randomized Controlled Trial Examining Motivation and Cognition in Stroke Patients
Brief Title: Ready, Set, Goal: Motivation and Cognition in Stroke Patients
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Richard H. Swartz, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 001
Record Dates: First submitted 2018-02-12; First posted 2018-04-27 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Stroke, Ischemic
Keywords: Cognition; Apathy
MeSH Terms: conditions — Ischemic Stroke; Lethargy

STUDY DESIGN:
Intervention Model Description: The study is a single-blind randomized controlled trial. It employs a mixed design, with a between-subjects (instruction type: goal-setting or standard instructions) and a within subjects (pre- and post-instruction manipulation) variable. Seventy-two stroke patients will undergo baseline cognitive testing to assess their verbal ability, learning, memory, attention, visuospatial ability, and exective functioning, with standardized instructions. After completing baseline testing and ratings of apathy (AES), depression (CES-D), anxiety, motivation, and fatigue, participants (N = 72) will either be assigned to the standardized instruction condition (n = 30) or the goal-setting instruction condition (n = 30).
Who Masked: Participant
Masking Description: Participants will not be told which group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Instructions (Placebo Comparator): Participants will receive standard instructions for cognitive tasks.
  Interventions: Behavioral: Standard Instructions
- Goal Setting Instructions (Experimental): Participants will receive goal-setting instructions for cognitive tasks.
  Interventions: Behavioral: Goal-Setting Instructions; Behavioral: Standard Instructions

INTERVENTIONS:
Behavioral: Goal-Setting Instructions — In the goal-setting instruction condition, participants will be asked to increase their performance by 20% from the previous similar test (e.g., "On this task, you generated 10 words when I asked you to name as many words as you could that start with the letter 'F.' Now, I want you to aim to generate at least 12 words for the letter 'F'.")
  Arms: Goal Setting Instructions
Behavioral: Standard Instructions — Participants in this group will receive the standardized instructions for completing the tests, as outlined in the test appendices.

SUMMARY:
Apathy is a syndrome of reduced motivation, characterized by diminished goal-directed behaviours (e.g., lack of effort), decreased goal-oriented cognitions (e.g., lack of interest) and blunted affect. Apathy is present in 20-50% of individuals after experiencing a stroke. Despite the detrimental impact of reduced goal-directed behaviours and cognitions on activities of daily living and cognition in stroke patients, interventions for increasing motivation (reducing apathy) have yet to be examined in this population. This study will examine the effect of goal-setting instructions on cognitive performance in stroke patients. The investigators hypothesize that in stroke patients, goal-setting instructions will improve cognitive performance relative to standard instructions. If goal-setting instructions are effective in improving cognitive performance, it may indicate that treatments targeting apathy could serve as a novel way to improve cognitive outcomes and enhance patient quality of life post-stroke.

DETAILED DESCRIPTION:
The study is a single-blind randomized controlled trial. It employs a mixed design, with a between-subjects variable (goal-setting instructions versus standardized instructions) and a within-subjects variable (pre-post instructional manipulation). It is a one-time intervention lasting 1-2 hours. Investigators plan to enroll 72 patients in this study. All participants will complete neuropsychological measures to assess their baseline performance. The baseline measures include Trial 1 of the CVLT-II Alternate Form, the Digit Span Test, Center for Epidemiologic Studies Depression Scale, Controlled Oral Word Association Test, Semantic Fluency Test, Apathy Evaluation Scale and Trail Making Test. After the baseline measures are completed, all participants will rate their level of motivation on a scale from 1 (extremely unmotivated) to 100 (extremely motivated), which will act as a pre-manipulation check measure, their level of fatigue on a scale from 1 (extremely not fatigued) to 100 (extremely fatigued), and their level of anxiety from 1 (extremely not anxious) to 100 (extremely anxious; 1 minute).

After completing the baseline measures and rating scales, half (n = 36) of the participants will be randomly assigned to the goal-setting instruction group ("goal-setting group"). Motivation will be enhanced by asking participants to perform 20% better than their previous performance on a similar task, and translating that into a number (e.g., "On this task, you generated 10 words when I asked you to name as many words as you could that start with the letter "F." Now, for the next letter, I want you to generate 12 words."). The remainder of the participants (n = 36) will be assigned to the "standard instruction group," where they will only receive the standardized instructions for completing the tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient attending Secondary Stroke Prevention Clinic
* Ischemic Stroke
* Presenting at least 3 months after stroke
* Modified Rankin Scale Score of at least 4
* Fluent in English

Exclusion Criteria:

* Marked aphasia
* Marked neglect
* Severe visual impairment
* Inability to complete 1 hour of cognitive testing in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Controlled Oral Word Association Task | 10 minutes
  Participant performance on Controlled Oral Word Association Task in goal setting instructions group compared to standard instruction group.

SECONDARY OUTCOMES:
Motivation Level | 2 minutes
  Participant self-reported motivation level in goal setting instruction group versus standard instruction group.
Cognitive Performance on Semantic Fluency Test | 10 minutes
  Participant performance on Semantic Fluency Test in goal setting instructions group compared to standard instruction group.
Digit Span Test | 10 minutes
  Participant performance on Digit Span Test in goal setting instructions group compared to standard instruction group.
California Verbal Learning Test-II | 10 minutes
  Participant performance on California Verbal Learning Test-II in goal setting instructions group compared to standard instruction group.
Trail Making Test | 10 minutes
  Participant performance on Trail Making Test in goal setting instructions group compared to standard instruction group.

CONTACTS AND LOCATIONS:
Overall Officials: Keera Fishman, B.Sc, Study Director — Sunnybrook Health Sciences Centre/ University of Ottawa
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available.

REFERENCES:
- [Background] Scheurich A, Fellgiebel A, Schermuly I, Bauer S, Wolfges R, Muller MJ. Experimental evidence for a motivational origin of cognitive impairment in major depression. Psychol Med. 2008 Feb;38(2):237-46. doi: 10.1017/S0033291707002206. Epub 2007 Nov 16. PMID 18005498
- [Background] REITAN RM. The relation of the trail making test to organic brain damage. J Consult Psychol. 1955 Oct;19(5):393-4. doi: 10.1037/h0044509. No abstract available. PMID 13263471
- [Background] Darvesh S, Leach L, Black SE, Kaplan E, Freedman M. The behavioural neurology assessment. Can J Neurol Sci. 2005 May;32(2):167-77. doi: 10.1017/s0317167100003930. PMID 16018151
- [Background] Delis, D. C., Kramer, J. H, Kaplan, E., & Ober, B. A. (2000). California Verbal Learning Test - Second edition. Adult version: Manual. San Antonio: Psychological Corporation.
- [Background] Benton, A. L., & Hamsher, K. (1976). Multilingual Aphasia Examination. Iowa City, Iowa: University of Iowa.
- [Background] Wechsler, D. (2008). Wechsler Adult Intelligence Scale-Fourth Edition. San Antonio, TX: Pearson.
- [Background] Marin RS. Apathy: a neuropsychiatric syndrome. J Neuropsychiatry Clin Neurosci. 1991 Summer;3(3):243-54. doi: 10.1176/jnp.3.3.243. PMID 1821241
- [Derived] Fishman KN, Ashbaugh AR, Swartz RH. Goal Setting Improves Cognitive Performance in a Randomized Trial of Chronic Stroke Survivors. Stroke. 2021 Jan;52(2):458-470. doi: 10.1161/STROKEAHA.120.032131. Epub 2021 Jan 20. PMID 33467876